CLINICAL TRIAL: NCT07325487
Title: Adaptive Deep Brain Stimulation Targeting the Interposed Nucleus to Treat Spinocerebellar Ataxia
Brief Title: Interposed Nucleus aDBS for Ataxia
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Florida (Other)
Collaborators: Raynor Cerebellum Project (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB202501191
Record Dates: First submitted 2026-01-05; First posted 2026-01-08 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2025-12

CONDITIONS: Spinocerebellar Ataxia (SCA); Spinocerebellar Ataxia Type 6
Keywords: SCA6; Spinocerebellar Ataxia; adaptive deep brain stimulation; aDBS; Spinocerebellar Ataxia Type 6; DBS; deep brain stimulation
MeSH Terms: conditions — Spinocerebellar Ataxias | interventions — Deep Brain Stimulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Adaptive Deep Brain Stimulation (aDBS) (Experimental): Participants will undergo surgical implantation of deep brain stimulation (DBS) leads targeting the motor interposed nucleus of the cerebellum. Approximately one month after implantation, participants will begin conventional DBS (cDBS) programming to identify optimal stimulation parameters, including amplitude, contact configuration, frequency, and pulse width, and to assess stimulation-related adverse effects and device function.
  Approximately nine months after implantation, stimulation settings will be transitioned to adaptive DBS (aDBS), in which stimulation amplitude is automatically adjusted based on recorded neural activity. Adaptive DBS will be used to evaluate the feasibility, safety, and tolerability of cerebellar aDBS.
  Clinical outcomes, symptoms, and potential side effects will be assessed throughout the study using participant self-reports, validated clinical rating scales, and wearable devices to collect movement and sleep data.
  Interventions: Device: Deep Brain Stimulation

INTERVENTIONS:
Device: Deep Brain Stimulation — This device will be surgically implanted into the interposed nucleus of the cerebellum.
  Other Names: Medtronic Percept

SUMMARY:
This is a single-center, open-label study designed to evaluate the feasibility, safety, and preliminary efficacy of cerebellar adaptive deep brain stimulation (aDBS) in adults with spinocerebellar ataxia type 6 (SCA6). A total of 5 participants will be enrolled.

Participants will undergo surgical implantation of deep brain stimulation (DBS) leads targeting the motor interposed nucleus of the cerebellum. The leads will be connected to one or two implantable pulse generators capable of delivering stimulation to deep brain structures and recording neural activity.

Participants will complete up to 18 in-person study visits over a 24-month follow-up period. During these visits, neural signals will be recorded under varying behavioral tasks and stimulation conditions.

Early study visits will be used to identify optimal stimulation parameters and neural biomarkers associated with disease state. These biomarkers will subsequently be used to implement adaptive DBS, in which stimulation amplitude is automatically adjusted in response to recorded neural activity.

Study outcomes will include assessments of safety and feasibility of cerebellar aDBS, as well as preliminary evaluation of its effects on clinical measures.

ELIGIBILITY:
Inclusion Criteria:

* A diagnosis of SCA6 by a movement disorders specialist following established criteria recommended by the Movement Disorders Society
* A positive genetic test for SCA6
* A total score ≥ 8 on the Scale of the Assessment and Rating of Ataxia (SARA) rating scale
* Ability to walk with or without support (score <8 on the 'gait' subsection of the SARA rating scale)
* Age ≥ 21 years and <89 years
* Ability to give informed consent for the study
* Ability to understand the study protocol

Exclusion Criteria:

* Inability or unwillingness to comply with the study protocol
* History of previously implanted neurostimulators, pacemakers, defibrillators, or metallic head implants
* Severe cognitive impairment or dementia, defined as a score <21 on the Montreal Cognitive Assessment (MOCA)
* Evidence of ataxia due to other etiologies, including but not limited to:

  * Genetic/inherited disorders other than SCA6
  * Acquired causes: traumatic brain injury, multiple sclerosis, paraneoplastic cerebellar degeneration, infections or post-infectious cerebellitis, autoimmune ataxias (e.g., anti-GAD, gluten ataxia)
  * Toxic/metabolic causes: alcoholic cerebellar degeneration, vitamin deficiencies
  * Structural, vascular, or neoplastic causes: cerebellar stroke, tumors, congenital malformations
  * Suspected multiple system atrophy-cerebellar type (MSA-C)
* Presence of active and untreated psychiatric illness, severe depression (Beck Depression Inventory ≥ 21), or personality disorder at the discretion of the study team
* Coagulopathy, uncontrolled epilepsy, or other medical conditions that are considered to place the patient at elevated risk for surgical complications
* Presence of a concomitant medical condition that, in the investigator's opinion, may interfere with the study participation or gait/balance, for example, severe arthritis
* Requirement of diathermy, electroconvulsive therapy, or transcranial magnetic stimulation
* Pregnancy or lactation
* Active suicidal ideation, defined as a "Yes" response to questions #2-5 on the Columbia Suicide Severity Rating Scale, C-SSRS
* Refractory epilepsy

Ages: 21 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Estimated)
Dates: Start 2026-03 (Estimated); Primary Completion 2031-03 (Estimated); Study Completion 2031-03 (Estimated)

PRIMARY OUTCOMES:
The identification of a physiological signal to use as the aDBS feedback signal | From baseline through study completion, about 2 years.
  Local field potentials (LFP) will be recorded in the clinic as well as chronically at home. These recordings will be analyzed to identify electrophysiological markers of disease states and therapeutic effects.
The incidence of unexpected adverse events and serious adverse events with aDBS compared to baseline | From baseline through study completion, about 2 years.
  Adverse events are monitored the entire time subject is enrolled in study. Unexpected and serious adverse events from baseline through study completion, about 2 years, is a primary endpoint.

SECONDARY OUTCOMES:
The Upright Balance Assessment measured by force plate parameters | From baseline through study completion, about 2 years.
  The Upright Balance Assessment is designed to evaluate walking and balance.
The Scale for the Assessment and Rating of Ataxia (SARA) | From baseline through study completion, about 2 years.
  The Scale for the Assessment and Rating of Ataxia (SARA) is an 8-item performance based scale used to determine the severity of ataxia. Scoring ranges from 0 to 40, with a higher score indicating greater ataxia severity.
The Patient-Reported Outcome Measure of Ataxia (PROM-Ataxia) | From baseline through study completion, about 2 years.
  The Patient-Reported Outcome Measure of Ataxia (PROM-Ataxia) is a 70-item scale divided into three domains of patient experiences assessing physical function, activities of daily living (ADL), and mental health. Scores range from 0 to 280, with a higher score indicating more severe symptoms and poorer quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Coralie de Hemptinne, PhD, Principal Investigator — University of Florida
Locations (1):
- Norman Fixel Institute for Neurological Diseases, Gainesville, Florida, United States

IPD SHARING:
Plan to Share IPD: No